CLINICAL TRIAL: NCT05213468
Title: Self-management of Chronic Pain Through the Use of the Digital Tool PainDrianer
Brief Title: Self-management of Chronic Pain Though E-health
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A change in patient population at the clinical trial site has occurred due to the pandemic, resulting in too few patients for the physiotherapy program to conduct the study.
Sponsor: PainDrainer AB (Industry)
Collaborators: Skane University Hospital (Other); Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUS-S1
Record Dates: First submitted 2022-01-05; First posted 2022-01-28 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Chronic Pain
Keywords: self management; e-health; health tech; Digital Pain-Management Tool
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Parallel study, single blinded
Who Masked: Care Provider
Masking Description: Parallel study, single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self management app as add on to standard care (Experimental): PainDrainerTM App as add on to standard treatment at the physiotherapy program at the clinic PainDrainer software application: PainDrainerTM app (version 1.1.19c). ' The PainDrainer app is an investigational device, intended as a digital aid for the self-management of chronic pain for use by adults without supervision by healthcare professionals in a home setting.
  Interventions: Device: PainDrainerTM
- Standard of care (No Intervention): Treatment as usual, standard treatment of care at the physiotherapy program at the clinic

INTERVENTIONS:
Device: PainDrainerTM — Self management digital tool for chronic pain
  Arms: Self management app as add on to standard care

SUMMARY:
The investigators aim to validate if a digital tool for increased self-management of chronic pain can improve the quality of life for patients with chronic pain. The validation is based on the change in pain interference (Quality of life), pain intensity, physical functioning, depression, and anxiety based on self-reported information from baseline to study end.

DETAILED DESCRIPTION:
Chronic pain is today an increasing health problem in both Europe and US, with an estimation of about 90 million people affected in Europe and 100 million people in US, or 20-30% of the adult population around the world. Chronic pain is defined as a condition that lasts for at least three to six months, after the normal healing period of an injury. Medical interventions offered in clinics around the globe are unfortunately not giving the results needed to give back the quality of life the patients had prior to the onset of the pain. The treatments offered today do sometimes reduce pain, but the effect is minor, and new treatment regimens are needed. Recent quality assurance registry measurements in Sweden has shown that patient taken part of multi modal treatment regimens, such as the acceptance and commitment therapy, (ACT) show that less then 40% of the patients have a decline in the pain level of 1 level on the VAS scale, 55% has no effect. The study objective is to evaluate how the use of a digital pain coach, based on artificial intelligence that improves the self-management of pain will decrease the pain interference and thereby increase QoL among chronic pain patients, as measured by PROMIS pain interference 6a. This study will compare the improvement of quality of life by a decrease in pain interference, measured by PROMIS, in patients who follow their traditional treatment plan provided by the Pain Clinic with the addition of using a web application for increased self management of pain. The theory behind the study and the development of the device is supported by previously known data, showing that self-management has an effect and is important to the treatment by helping patients to believe in their own capacity to control their pain.

The present investigation aims at exploring the effect of including digital tool as an add on to standard treatment and rehabilitation at the physiotherapy program at the clinic and will measure the effect it has on:

1. Decreased pain interference
2. Improved management of long-term pain and its consequences. Hence self management of pain
3. Increased function in daily life with the best possible activity and participation level
4. Improved experience of health-related quality of life
5. Decreased pain experience

ELIGIBILITY:
Inclusion Criteria:

* Have a pain condition that requires analysis and rehabilitation at a specialist clinic
* >18 years of age
* Be medically investigated, with adequate pharmacological treatment, and do not have any other medical examination or ongoing illness that hinders participation in the physiotherapy program at VO Neurosurgery and Pain rehabilitation, Skåne University Hospital, Lund
* Meet the criteria for inclusion in the physiotherapy program: Have a chronic (> 3 months) state of pain with local, regional or spread location, where the pain is judged to be reduced by physiotherapeutic measures
* Being included in the physiotherapy program, at VO Neurosurgery and Pain rehabilitation, Skåne University Hospital, Lund
* Have the knowledge and proficiency to use a smart phone, tablet or computer

Exclusion Criteria:

* Severe or acute psychiatric illness, severe anxiety or depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Pain interference | 6 and 12 weeks from baseline
  Change from baseline in pain interference (QoL), measured by PROMIS Pain Interference 4a . Measure of the amount of interference pain causes in life; range 4-20; higher is worse

SECONDARY OUTCOMES:
Pain severity | 6 and 12 weeks from baseline
  Change from Baseline in the 7 day average pain intensity. Measured by NRS using Pain Intensity Numerical Rating Scale (NRS) (0=no pain, 10=pain as bad as you can imagine)
Physical function | 6 and 12 weeks from baseline
  Change from baseline in physical function, measured with Patient-Reported Outcomes Measurement Information System (PROMIS) Physical function 4a.
  Measure of the impact of a condition on physical function; range 4-20; Raw scores range from 4-20 with higher scores represent better functioning.
Depression | 6 and 12 weeks from baseline
  Change from Baseline measured with Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Depression 4a.
  Measures the extent to which patients experience depressive symptoms over the past 7 days. Raw scores range from 4-20 with higher scores represent worse symptomatology.
Anxiety | 6 and 12 weeks from baseline
  Change from Baseline measured with Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress - Anxiety 4a.
  Measures the extent to which patients experience anxiety symptoms over the past 7 days. Raw scores range from 4-20 higher scores represent worse symptomatology.
Fatigue | 6 and 12 weeks from baseline
  Change from Baseline measured with Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue 4a Measures the extent to which patients experience fatigue symptoms over the past 7 days. Raw scores range from 4-20 with higher scores represent worse symptomatology.
Sleep disturbance | 6 and 12 weeks from baseline
  Change from Baseline measured with Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep disturbance 4a Measures the extent to which patients experience Sleep disturbance over the past 7 days. Raw scores range from 4-20 with higher scores represent worse symptomatology.
Ability to Participate in Social Roles and Activities | 6 and 12 weeks from baseline
  Change from Baseline measured with Patient-Reported Outcomes Measurement Information System (PROMIS) Ability to Participate in Social Roles and Activities 4a. Measures the extent to which patients ability to participate in social roles and activities over the past 7 days. Raw scores range from 4-20 with higher scores represent better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Rivano Fischer, Clin.Psy.D, Principal Investigator — VO Neurosurgery and Pain rehabilitation, Skåne University Hospital, Lund
Locations (1):
- VO Neurokirurgi och Smärtrehabilitering Skånes universitetssjukhus, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No